CLINICAL TRIAL: NCT04387864
Title: The Effect of Adding Whole-Body Vibration Exercises to Home Exercise Program on Muscle Strength in Patients With Postpolio Syndrome
Brief Title: Whole Body Vibration on Muscle Strength in Patients With Postpolio Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015/1262
Record Dates: First submitted 2020-05-10; First posted 2020-05-14 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Postpolio Syndrome
Keywords: postpolio syndrome; whole body vibration; exercises; muscle strength; poliomiyelitis
MeSH Terms: conditions — Postpoliomyelitis Syndrome; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole-body Vibration Exercise Group (Experimental): The patients in the WBV exercise group underwent WBV exercise sessions 2 days a week (72 hours in between) for a total of 6 weeks. Each exercise session was performed under the supervision of a physician.
  The patients received support from both hands on the WBV platform and both knees were positioned statically at 40-60 degree flexion (high squat position). All patients stood on the platform with sports socks (without shoes) to avoid the shoes absorbing vibration. Vibration was given by a Power Plate® device where a three-plane oscillation occurs (most vertical, Z axis). In all vibrations, 30 Hz frequency and 2 mm amplitude (low amplitude) were used. The vibration time was set to be 30 seconds in the first two weeks, 45 seconds in the next two weeks and 60 seconds in the last two weeks. The repetition of vibration was increased by 1 repetition every week, starting with 5, and 10 repetitions were given in the last week. A 1-minute rest period was given between each repetition.
  Interventions: Device: Whole-body Vibration Device
- Home Exercise Group (No Intervention): The home program, which included isometric and isotonic exercises, was followed at home for 6 weeks. Three sets of quadriceps setting as 5 repetitions, 5-second contractions, and three sets of isotonic quadriceps exercise in seating position with weights as 12 repetitions were administered to be performed two days a week. While the patients included in the study group came for TVT exercise two days a week, the patients in the control group performed quadriceps setting exercises also on those days. The patients were invited to the physician follow-up on Wednesday every week for motivation and follow-up. The patients were asked to write their complaints during and after the exercise, if any. In addition, they were asked to note the number of repetitions and sets of their exercises on exercise booklets prepared for the patient.

INTERVENTIONS:
Device: Whole-body Vibration Device — Power Plate® (pro5TM; Power Plate North America, Inc., Northbrook, IL, USA)
  Arms: Whole-body Vibration Exercise Group

SUMMARY:
Post-polio syndrome (PPS) is a neurological disease that affects polio survivors at least 15 years after the initial polio infection. PPS is characterized by new neurological deficiencies after a period of neurological stability, especially at least 1 decade after the initial infection. PPS may manifest as new, persistent, and progressive muscle weakness, atrophy, limb fatigability, myalgia, arthralgia, and dysphagia, but also as generalized fatigue, which typically has a considerable impact on the patients' quality of life. Whole body vibration (WBV) has become a popular form of exercise therapy especially among elderly individuals, in past decades. This training method is performed by standing on a vibrating platform which is supposed to activate muscle contractions. WBV has been studied in neurologic populations with stroke, Parkinson's disease, cerebral palsy, incomplete spinal cord injury, and multiple sclerosis.Our aim was to investigate the effectiveness of whole-body vibration (WBV) exercises performed with home exercise program and patient education in patients with postpolio syndrome (PPS) on muscle strength, fatigue, quality of life and laboratory parameters by comparing them with home exercise program and patient education alone.

DETAILED DESCRIPTION:
Post-polio syndrome (PPS) is a neurological disease that affects polio survivors at least 15 years after the initial polio infection. The description of PPS is attributed to Jean-Martin Charcot in 1875 but was only widely recognized in the early 1980s [1].

PPS is characterized by new neurological deficiencies after a period of neurological stability, especially at least 1 decade after the initial infection. PPS may manifest as new, persistent, and progressive muscle weakness, atrophy, limb fatigability, myalgia, arthralgia, and dysphagia, but also as generalized fatigue, which typically has a considerable impact on the patients' quality of life. The estimates of the percentage of polio patients affected by PPS are inconsistent, varying between 20 and 85% depending on the diagnostic criteria applied [1].

Despite its prevalence, post-polio syndrome remains surprisingly under-researched. People with PPS generally have fewer options for exercise because it may exacerbate PPS symptoms such as pain, fatigue, and muscle weakness [2].

The pathophysiological framework relating to the genesis of PPS is based on the theory of super training, considering that shortly after an episode of acute poliomyelitis, the remaining motor neurons increase the number of sprouts for the reinnervation of muscle fibers after they have been denervated. About two to three decades after the acute episode, there is a tendency to overload this system, that can be accelerated depending on individual factors especially the activities and exercises carried out that promote overuse of the affected muscles. In this case of overuse and super training, an intense metabolic demand in the residual motor units occurs, which then triggers a process of secondary neuronal death, and active inflammatory process is present in the spinal cord with increased level of cytokines in the cerebrospinal fluid but without any convincing evidence of viral reactivation. Another hypothesis for the genesis of PPS is that it results from an autoimmune disorder, a theory that is reinforced by the presence of anti-neurofilament antibodies in the cerebrospinal fluid [1, 3, 4].

There is an ongoing process of denervation and reinnervation in the muscle fibers of motor units that survived in PPS patients. Excessive physical activity accelerates the loss of motor units. Therefore, it is very important to plan the exercise so as not to cause additional harmful effects on the integrity of the muscle and survived motor units, to ensure maximal improvement and to prevent overload.

In Cochrane review published in 2015, Koopman et al. reported that data on the effectiveness of muscle strengthening in PPS was controversial. In two studies, it was stated that strengthening thumb muscles and applying static magnetic field were reliable and effective, they increased muscle strength, but their effect on functional limitation was unknown. There is not any available data on the effectiveness of exercise for major muscle groups [5].

Whole body vibration (WBV) has become a popular form of exercise therapy especially among elderly individuals, in past decades. This training method is performed by standing on a vibrating platform which is supposed to activate muscle contractions. WBV has been studied in neurologic populations with stroke, Parkinson's disease, cerebral palsy, incomplete spinal cord injury, and multiple sclerosis, with del Pozo-Cruz et al. conducting a systematic review presenting varying results pertaining to impairments, activity limitations, and health-related quality of life. Limited data is available about the WBV in patients with polio syndrome [6].

ELIGIBILITY:
Inclusion Criteria:

* having a knee flexion and extension
* muscle strength of >3/5 according to the manual muscle strength evaluation on the healthy lower extremity
* walking 300 meters alone with or without an assistive device

Exclusion Criteria:

* epilepsy
* the presence of a cardiac pacemaker
* a history of previous hip or knee prosthesis
* bleeding diathesis
* uncontrolled diabetes
* obesity (BMI≥30 kg/m2)
* pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-03-25 (Actual)

PRIMARY OUTCOMES:
Muscle Strength Assessment | 6 weeks
  In our study, knee extensor and flexor muscle strengths were measured with a CybexTM (Humac) Norm 350 (Cybex Norm, Lumex Inc., Ronkonkoma, New York, USA) computed isokinetic dynamometer device. The tests were performed by an exercise physiologist with nearly 20 years of experience in isokinetic measurement and rehabilitation. It was ensured that the patients were not fasting and went to the toilet before the muscle test. Usually, the same time of day was preferred and maximum three patients were assessed per day. Each patient underwent a total of two measurements before and after the study. Care was exerted to ensure that the measurements were performed 48 hours after the end of the exercise.

SECONDARY OUTCOMES:
Fatigue Severity Scale (FSS) | 6 weeks
  It is a scale developed to measure the severity of fatigue. It is a valid and reliable assessment scale for evaluating PPS-related fatigue. The scale questions the severity of fatigue within the last month. The scale consists of 9 items and each item is rated on a 7-point scale. High scores indicate fatigue, while a score of ≥28 points indicate the presence of fatigue
Fatigue Impact Scale (FIS) | 6 weeks
  The fatigue impact scale was developed to evaluate fatigue symptoms in chronic diseases or conditions. It consists of forty items. It assesses the effects of fatigue on 3 dimensions of daily life activities: cognitive function, physical function and psychosocial function. Concentration concerns, memory, thinking and organization of though are questioned in cognitive function. Strength, coordination, effort and motivation are questioned in physical function. The effects of fatigue on workload and social isolation are questioned in psychosocial function. The scale questions the last 1 month. Each question is rated between 0 (no problem) and 4 (maximum problem). The highest score is 160 points
Nottingham Health Profile (NSP) | 6 weeks
  Health-related quality of life was assessed by the Nottingham Health Profile (NSP) scale, which the participants assessed themselves.
  In this scale, patients are asked to answer the questions as yes and no. It includes a total of 38 items and consists of 6 dimensions. Pain and physical activity are questioned in 8 items, sleep in 5 items, fatigue in 3 items, social isolation in 5 items, and emotional reaction are questioned in 9 items. The weighted score of that item is given to each yes answer given by the patients and 0 points to each no answer. In each dimension, points are calculated separately. Each category takes a value between 0-100. Thus, health profile score is obtained
Muscle Damage Assessment | 6 weeks
  Exercise is known to cause muscle damage to varying extents. Muscle damage is a condition that causes exhaustion, loss of function, weakness and pain in muscles after unfamiliar and heavy exercises. In our study, the levels of creatine kinase (CK), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) were studied in the serum of the patients before and 48 hours after the exercise program ended to evaluate muscle damage.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşegül Ketenci, Prof, Principal Investigator — Istanbul University
Locations (1):
- Istanbul Faculty of Medicine, Istanbul University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Li Hi Shing S, Chipika RH, Finegan E, Murray D, Hardiman O, Bede P. Post-polio Syndrome: More Than Just a Lower Motor Neuron Disease. Front Neurol. 2019 Jul 16;10:773. doi: 10.3389/fneur.2019.00773. eCollection 2019. PMID 31379723
- [Result] Bruno, R.L., The polio paradox: What you need to know. 2009: Grand Central Publishing.
- [Result] Ghelman R, Akiyama IY, de Souza VT, Falcao J, Orgolini V, Hosomi JK, Quadros AAJ, Oliveira ASB. A twelve-week, four-arm, randomized, double-blind, placebo-controlled, phase 2 prospective clinical trial to evaluate the efficacy and safety of an anthroposophic multimodal treatment on chronic pain in outpatients with postpolio syndrome. Brain Behav. 2020 Apr;10(4):e01590. doi: 10.1002/brb3.1590. Epub 2020 Mar 11. PMID 32162497
- [Result] Lo JK, Robinson LR. Postpolio syndrome and the late effects of poliomyelitis. Part 1. pathogenesis, biomechanical considerations, diagnosis, and investigations. Muscle Nerve. 2018 Dec;58(6):751-759. doi: 10.1002/mus.26168. Epub 2018 Aug 22. PMID 29752819
- [Result] Koopman FS, Beelen A, Gilhus NE, de Visser M, Nollet F. Treatment for postpolio syndrome. Cochrane Database Syst Rev. 2015 May 18;2015(5):CD007818. doi: 10.1002/14651858.CD007818.pub3. PMID 25984923
- [Result] del Pozo-Cruz B, Adsuar JC, Parraca JA, del Pozo-Cruz J, Olivares PR, Gusi N. Using whole-body vibration training in patients affected with common neurological diseases: a systematic literature review. J Altern Complement Med. 2012 Jan;18(1):29-41. doi: 10.1089/acm.2010.0691. Epub 2012 Jan 10. PMID 22233167
- [Result] Koopman FS, Brehm MA, Heerkens YF, Nollet F, Beelen A. Measuring fatigue in polio survivors: content comparison and reliability of the Fatigue Severity Scale and the Checklist Individual Strength. J Rehabil Med. 2014 Sep;46(8):761-7. doi: 10.2340/16501977-1838. PMID 24941350
- [Result] Fisk JD, Ritvo PG, Ross L, Haase DA, Marrie TJ, Schlech WF. Measuring the functional impact of fatigue: initial validation of the fatigue impact scale. Clin Infect Dis. 1994 Jan;18 Suppl 1:S79-83. doi: 10.1093/clinids/18.supplement_1.s79. PMID 8148458
- [Result] Oncu J, Atamaz F, Durmaz B, On A. Psychometric properties of fatigue severity and fatigue impact scales in postpolio patients. Int J Rehabil Res. 2013 Dec;36(4):339-45. doi: 10.1097/MRR.0b013e3283646b56. PMID 23903028
- [Result] Nollet F, Beelen A, Prins MH, de Visser M, Sargeant AJ, Lankhorst GJ, de Jong BA. Disability and functional assessment in former polio patients with and without postpolio syndrome. Arch Phys Med Rehabil. 1999 Feb;80(2):136-43. doi: 10.1016/s0003-9993(99)90110-7. PMID 10025486